CLINICAL TRIAL: NCT01716663
Title: CARTO® 3 System and Real Time Intracardiac Ultrasound for Ablation of Drug Refractory Recurrent Symptomatic Paroxysmal AF: Acute Procedural Outcomes Study
Brief Title: CARTO® 3 System and Real Time Intracardiac Ultrasound
Acronym: IUAF
Status: Completed | Type: Observational
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IUAF
Record Dates: First submitted 2012-10-19; First posted 2012-10-30 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Atrial Fibrillation; Paroxysmal AF
Keywords: Symptomatic paroxysmal; Atrial fibrillation; Observational; Acute procedural outcomes; Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental: Catheter Ablation: These patients have drug refractory recurrent symptomatic paroxysmal AF, are 18 years and older, and are able and willing to provide written informed consent to participate in the study and comply with study requirements.
  Interventions: Device: Catheter Ablation

INTERVENTIONS:
Device: Catheter Ablation — NAVISTAR® THERMOCOOL® SF Catheter with the CARTO® 3 System and the SOUNDSTAR® Ultrasound Catheter (with the CARTOSOUND® Software Module)
  Other Names: CARTO® 3 System and Real Time Intracardiac Ultrasound

SUMMARY:
This is a prospective, multicenter, non-randomized observational study of subjects 18 years and older undergoing RF ablation with drug refractory recurrent symptomatic paroxysmal Atrial Fibrillation (AF).

DETAILED DESCRIPTION:
This study is purposed to measure "real world" acute procedural outcomes (procedural efficiency and acute safety) associated with use of the CARTO® 3 System and real time intracardiac ultrasound in a clinical setting in subjects with drug refractory recurrent symptomatic paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

* Drug refractory, recurrent symptomatic paroxysmal AF
* Age 18 years or older
* Patients able and willing to provide written informed consent to participate in the study and comply with study requirements

Exclusion Criteria:

* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Previous ablation for atrial fibrillation
* AF episodes that last longer than 30 days
* Uncontrolled heart failure, or NYHA Class III or IV heart failure
* Documented intra-atrial thrombus or other abnormality on pre-ablation imaging
* Contraindication to anticoagulation
* Stroke, cardiac surgery, unstable angina, myocardial infarction or percutaneous coronary intervention within the past 3 months
* Awaiting cardiac transplantation
* Heart disease for which corrective surgery is anticipated within 6 months
* Enrollment in other investigational drug or device study
* Subjects unwilling to comply with protocol or follow-up requirements
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years and older with drug refractory recurrent symptomatic paroxysmal AF
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Usman Siddiqui, MD, Principal Investigator — Osceola Regional Medical Center; Mathew Hutchinson, MD, Principal Investigator — University of Pennsylvania; Andy Tran, MD, Principal Investigator — Scottsdale Healthcare Research; Saumil Oza, MD, Principal Investigator — East Coast Institute for Research LLC, St. Vincent's Ambulatory Care, Inc.; Robert Fishel, MD, Principal Investigator — JFK Medical Center; Vijendra Swarup, MD, Principal Investigator — AZ Heart Rhythm Research Center; Mohit Rastogi, MD, Principal Investigator — Washington Adventist Hospital CCVR; Brett Gidney, MD, Principal Investigator — Santa Barbara Cottage Hospital; John Scherschel, MD, Principal Investigator — University of Nebraska; Dilip Mathew, MD, Principal Investigator — Pepin Heart Hospital; William Sauer, MD, Principal Investigator — University of Colorado, Denver; Marcie Berger, MD, Principal Investigator — Medical College of Wisconsin; Khawaja Baig, MD, Principal Investigator — Kettering Medical Center; Farhat Khairallah, MD, Principal Investigator — Tallahassee Research Institute; David Fitzgerald, MD, Principal Investigator — Scott & White Memorial Hospital; Gopi Dandamudi, MD, Principal Investigator — Geisinger Heart Institute; Ahmad Abdul-Karim, MD, Principal Investigator — Provena St. Joseph Medical Center; Douglas Esberg, MD, Principal Investigator — Main Line Health; Scott Burke, MD, Principal Investigator — St. Mary's Medical Center; Gregory Jones, MD, Principal Investigator — Wellmont CVA Heart Institute; Tapan Rami, MD, Principal Investigator — The Methodist Hospital Research Institute; Salem Sayar, MD, Principal Investigator — Northeast Georgia Heart Center, PC; Gunjan Shukla, MD, Principal Investigator — Hackensack Meridian Health; Philip Gentlesk, MD, Principal Investigator — Sentara Norfolk General Hospital; Asim Yunus, MD, Principal Investigator — Michigan CardioVascular Institute; Scott Reich, MD, Principal Investigator — Northeast Baptist Hospital
Locations (26):
- United States (26):
  - AZ Heart Rhythm Research Center, Phoenix, Arizona
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - University of Colorado Denver, Aurora, Colorado
  - JFK Medical Center, Atlantis, Florida
  - East Coast Institute for Research, LLC. St. Vincent's Ambulatory Care, Inc., Jacksonville, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Pepin Heart Hospital, Tampa, Florida
  - Northeast Georgia Heart Center, PC, Gainsville, Georgia
  - Provena St. Joseph Medical Center, Joliet, Illinois
  - Washington Adventist Hospital CCVR, Takoma Park, Maryland
  - Michigan CardioVascular Institute, Saginaw, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Kettering Medical Center, Kettering, Ohio
  - St. Mary Medical Center, Newtown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Heart Institute, Wilkes-Barre, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas
  - Northeast Baptist Hospital, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: Catheter Ablation
Started | 234 (Enrolled = signed informed consent and met eligibility requirements)
Safety | 230 (Enrolled patients who had a study device inserted.)
Completed | 228 (Effectiveness population = enrolled and treated (study device inserted and RF energy applied))
Not Completed | 6
Not completed — Withdrawn prior to procedure | 4
Not completed — Treated with non-study catheter | 2

BASELINE CHARACTERISTICS:
Population: Enrolled
Arm/Group | Experimental: Catheter Ablation
Number analyzed (Participants) | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 120
  >=65 years | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 230
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 223
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Fluoroscopy Time
Description: The fluoroscopy time will be measured for each phase (access, mapping, ablation, and validation) of the procedure and summed to derive the total.
Time Frame: Day 0
Population: Those patients with non-missing fluoroscopy time.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Experimental: Catheter Ablation
Number analyzed (Participants) | 221
minutes | 28.3 (29.71)

2. Secondary Outcome: Total Procedure Time
Description: The procedure time will be measured for each phase (access, mapping, ablation, and validation) of the procedure and summed to derive the total.
Time Frame: Day 0
Population: The number of patients with non-missing procedure time data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Experimental: Catheter Ablation
Number analyzed (Participants) | 225
minutes | 150.2 (76.32)

3. Secondary Outcome: Acute Procedural Success
Description: Acute success will be defined as confirmation of pulmonary vein isolation by entrance block, exit block, and/or periostial block of all targeted pulmonary veins.
Time Frame: Day 0
Population: Acute effectiveness and efficiency cohort
Measure: Number; unit: participants
Arm/Group | Experimental: Catheter Ablation
Number analyzed (Participants) | 228
participants | 226

4. Secondary Outcome: Mean Number of Radiofrequency (RF) Applications
Description: RF application is defined as the number of times RF energy is delivered during the procedure.
Time Frame: Day 0
Population: Patients with non-missing RF application values
Measure: Mean (Standard Deviation); unit: number of applications
Arm/Group | Experimental: Catheter Ablation
Number analyzed (Participants) | 227
number of applications | 54.2 (43.95)

5. Secondary Outcome: Total Radiofrequency (RF) Time
Description: Total RF time is defined as the total time RF is delivered during the procedure.
Time Frame: Day 0
Population: Patients with non-missing RF application time.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Experimental: Catheter Ablation
Number analyzed (Participants) | 227
minutes | 104.7 (57.64)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Experimental: Catheter Ablation
Serious Adverse Events (participants affected / at risk) | 22/230
Other Adverse Events (participants affected / at risk) | 13/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Catheter Ablation (N=230)
atrial fibrillation (Cardiac disorders) | 1
atrial flutter (Cardiac disorders) | 1
atrioventricular block (Cardiac disorders) | 1
cardiac failure congestive (Cardiac disorders) | 2
pericardial effusion/tamponade (Cardiac disorders) | 3
pericarditis (Cardiac disorders) | 3
vertigo positional (Ear and labyrinth disorders) | 1
chest pain (General disorders) | 1
puncture site hemorrhage (General disorders) | 1
pneumonia (Infections and infestations) | 1
post procedural hematoma (Injury, poisoning and procedural complications) | 1
vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2
cardiac telemetry abnormal (Investigations) | 1
fluid overload (Metabolism and nutrition disorders) | 1
migraine (Nervous system disorders) | 1
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Catheter Ablation (N=230)
atrial fibrillation (Cardiac disorders) | 7
pericarditis (Cardiac disorders) | 3
pyrexia (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present, or publish trial results after the trial is completed. Please contact Biosense Webster for additional information.